CLINICAL TRIAL: NCT01732978
Title: Are Parents Privileged Listeners Their Baby ?
Acronym: BABIES_CRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1208093
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Newborn
Keywords: Crying record; Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Babies (Other): Any child born in the University Hospital of Saint Etienne (inborn) whatever its term birth, hospitalized in a neonatal unit at the time of registration (after 37 weeks of gestation for preterm infants) or maternity
  Interventions: Behavioral: Crying record

INTERVENTIONS:
Behavioral: Crying record — Recording spontaneous crying is as soon as possible after birth. Crying is recorded twice during the first week of life.
  Listening tests:
  Tests will be conducted playbacks with the father and mother separately, and with a staff

SUMMARY:
The crying baby is a sound signal including information relating to this individual identity or related to its physiological or motivational state.

The objective of the study is to determine the implementation of the recognition of individual tone of the baby by his parents and acoustic modulation of the baby based on parental response.

The detailed study of the acoustic structure of crying and analysis of parental perception will determine the dynamics during the first weeks of life of this recognition, and the influence of factors such as parental presence, or breastfeeding .

For this study is organized in three stages: first, the recording of the baby's crying Secondly, a listening test parental soundtracks and third analysis of the acoustic structure of crying and parental response.

ELIGIBILITY:
Inclusion Criteria:

* born in the University Hospital of Saint Etienne (inborn) whatever its term birth

Exclusion Criteria:

* Congenital oropharyngeal tract preventing vocalization physiological newborn

Max Age: 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Crying recorded | Second day of life of the parent's child
  The acoustic structure of crying recorded the first days of life will be analyzed and aims to characterize an individual signature and the dynamic function of time of this structure.

SECONDARY OUTCOMES:
Biological correlation | Second day of life of parents' child
  The acoustic structure of crying will also be studied to establish a possible correlation with biological parameters baby

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MATHEVON, PhD, Study Chair — Jean Monnet University
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France